CLINICAL TRIAL: NCT05169242
Title: A Double Blinded Randomized Controlled Trial on Prophylactic Clipping to Prevent Post-polypectomy Bleeding After Colonoscopy in Direct Oral Anticoagulant Users
Brief Title: A Trial on Prophylactic Clipping to Prevent Post-polypectomy Bleeding After Colonoscopy in Direct Oral Anticoagulant Users
Acronym: PROCLIP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Louis Ho Shing Lau, Resident Specialist, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2021.381
Record Dates: First submitted 2021-09-09; First posted 2021-12-23 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Post Polypectomy Bleeding

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): In the intervention arm, one or more endoclips will be used to completely close the mucosal defect after polypectomy. Prophylactic clipping will be applied to all post-polypectomy sites. The total number of endoclips used will be recorded.
  Interventions: Procedure: Endoclip
- Control group (No Intervention): In the control arm, no endoclip will be applied to all post-polypectomy sites, with the exceptions of uncontrolled immediate PPB or pre-treatment in very large pedunculated polyps as specified above. The subjects with endoclips applied due to safety reasons will be included in the subsequent intention-to-treat analysis, but not the per-protocol analysis.

INTERVENTIONS:
Procedure: Endoclip — In the intervention arm, one or more endoclips will be used to completely close the mucosal defect after polypectomy. Prophylactic clipping will be applied to all post-polypectomy sites. The total number of endoclips used will be recorded.
  Arms: Intervention group

SUMMARY:
The investigators hypothesize that prophylactic clipping after colonoscopic polypectomy can reduce risk of delayed PPB among DOAC users. The investigators also hypothesize that pre-endoscopy drug level can predict the risk of hemorrhagic complications after the procedure.

DETAILED DESCRIPTION:
Despite the clinical benefit of colonoscopic polypectomy, post-polypectomy bleeding (PPB) occurs in up to 6.5% of patients. Current international guidelines classify polypectomy as one of the endoscopic procedures with high risk of hemorrhage.

Risk factors for PPB include advanced age, cardiovascular or renal diseases, large polyp size, pedunculated morphology, proximal location in right colon, and the use of antithrombotic medications. Among them, the use of oral anticoagulants such as warfarin and direct oral anticoagulants (DOAC) is associated with a substantially higher risk of PPB up to 13.7%.

While prophylactic clipping is often performed by endoscopists to reduce the PPB risk in clinical practice, the available evidence on its efficacy has been heterogenous and conflicting. A number of studies reported the efficacy of prophylactic clip closure after endoscopic resection to prevent PPB. On the contrary, several randomized trials did not demonstrate any significant benefit of prophylactic clipping. In recent meta-analyses, routine use of prophylactic clipping was not shown to decrease PPB risk, except in a subgroup of colonic lesion larger than 20mm and proximal to the hepatic flexure. However, the proportion of patients on oral anticoagulants was low (5.1%-26%) in the above studies, limiting the generalizability of results to this high-risk patient group. Our preliminary data involving >500 patients on oral anticoagulants showed a lower PPB risk in prophylactic clipping group among DOAC users.

Also, although the consensus is that DOAC users do not require routine drug level monitoring, studies have shown a positive correlation between plasma drug level and bleeding risks. In special circumstances, the measurement of anticoagulant effect would provide management guide, including patients with extreme body weight or renal impairment, imminent need of antidote reversal or before invasive surgical procedures. Diluted thrombin time and anti-factor Xa assays demonstrated a reasonable linear correlation with the plasma drug concentration, yet they are indirect tests. Specific DOAC drug level can be checked to provide direct measurement of anticoagulant effect. In the setting of elective invasive procedures, a pre-operative cutoff level (≦30 ng/mL) for dabigatran and rivaroxaban has been proposed. Patients undergoing interventions with high bleeding risks may benefit from drug level measurement by informing the operators to perform prophylactic measures to reduce hemorrhagic complications.

In this randomized controlled trial, we aim to evaluate the efficacy of prophylactic clipping in preventing PPB in colonoscopy among DOAC users. We also wish to investigate the correlation of pre-endoscopy DOAC drug level and the risk of hemorrhagic complications after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* They are active users of any DOAC
* They require elective colonoscopy for colorectal cancer screening, polyp surveillance, or investigation of symptoms such as anemia or past gastrointestinal bleeding
* Aged 18 years old or above;
* Written informed consent obtained.

Exclusion Criteria:

* Absolute contraindications to colonoscopy
* Any medical conditions precluding interruption of DOAC for procedure
* Any medical conditions requiring concomitant uninterrupted dual antiplatelet drugs (single antiplatelet drug users will not be excluded)
* Active gastrointestinal bleeding
* Clinically significant bleeding tendency (decompensated cirrhosis or severe thrombocytopenia)
* Severe renal impairment (defined as creatinine clearance < 15 ml/min)
* Pregnancy or lactation;
* Advanced comorbid conditions (defined as American Society of Anesthesiologists grade 4 or above)
* Unable to obtain informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 584 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2024-12-14 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinically significant delayed post-polypectomy bleeding | 2 years
  The primary endpoint is clinically significant delayed post-polypectomy bleeding.

SECONDARY OUTCOMES:
Overall delayed post-polypectomy bleeding rate and cardio-thrombotic event rate | 2 years
  Secondary endpoints are overall delayed post-polypectomy bleeding rate, cardio-thrombotic event rate within 30 days after procedure and pre-endoscopy DOAC drug levels. Overall delayed post-polypectomy bleeding is defined as occurrence of any gastrointestinal bleeding within 30 days after index colonoscopy (including those not fulfilling the criteria of primary endpoint). Cardio-thrombotic events are defined according to the Antithrombotic Trialists' criteria (non-fatal myocardial infarction, non-fatal stroke, or death from cardiovascular cause). [44] The baseline and trough DOAC drug levels measured before colonoscopy would also be analyzed and correlated with clinical bleeding or thrombotic events.

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Shatin, New Territories, Hong Kong

IPD SHARING:
Plan to Share IPD: No